CLINICAL TRIAL: NCT05580341
Title: A Phase III, Randomized, Blinded, Positive-controlled Study to Compare the Immunogenicity of Zerun 9-valent Human Papillomarivus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Pichia Pastoris) in Healthy Female Subjects Aged 16-26 Years.
Brief Title: Phase III Study Comparing the Immunogenicity of 9-valent HPV Recombinant Vaccine and Gardasil-9
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 312-HPV-2002
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cervical Cancer; Genital Wart; CIN; VIN; Papillomavirus Infections
Keywords: Human Papillomavirus; Papillomavirus Vaccines; Genital Warts; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zerun HPV-9 (Experimental): Subjects receive 3 doses of Zerun HPV-9 vaccine
  Interventions: Biological: Zerun HPV-9
- GARDASIL®9 (Active Comparator): Subjects receive 3 doses of GARDASIL®9
  Interventions: Biological: GARDASIL ®9

INTERVENTIONS:
Biological: Zerun HPV-9 — Zerun 9-valent Human Papillomarivus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Pichia Pastoris), 0.5mL, three doses, 0,2,6 months
  Arms: Zerun HPV-9
Biological: GARDASIL ®9 — GARDASIL®9 vaccine, 0.5mL, three doses, 0,2,6 months
  Arms: GARDASIL®9

SUMMARY:
This study will evaluate the immunogenicity and safety of Zerun 9-valent HPV recombinant vaccine in healthy female 16-26 years of age by comparing with GARDASIL®9.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female 16-26 years of age
* 16-17 years old subjects and their guardians able to provide legal identification; 18-26 years old subjects able to provide their legal identification;
* Able to understand (not illiterate) and sign the informed consent;
* Able to make a decision to participate in the clinical trial and the subject agrees to participate in the clinical trial;
* Women of child-bearing age (WOCBA): subjects must have a negative urine pregnancy test result, have used effective contraceptive measures within 2 weeks before enrollment, have no pregnancy plans, and agree to use adequate contraceptive precautions from enrollment to the 7th month (one month after full immunization).

Exclusion Criteria:

* Abnormal cervical cancer screen test results (ASC-US or worse), history of HPV infection, history of abnormal cervical biopsy results, or history of genital warts;
* Subjects with severe congenital malformations or that cause serious organ damage, developmental disorders, genetic defects, or severe malnutrition;
* Subjects have received a marketed HPV vaccine or participated in an HPV vaccine clinical trial, or participated in clinical trials of other vaccines within the past 6 months;
* Fever prior to vaccination (axillary body temperature ≥37.3℃);
* History of severe allergic reaction that required medical intervention (such as swelling of the mouth and throat, dyspnea, hypotension or shock, etc.);
* History of allergic to vaccine, or to any ingredient of vaccine (Aluminum phosphate adjuvant, sodium chloride, histidine, polysorbate 80),or history of severe adverse reaction
* History of epilepsy, psychosis, major depression requiring medication, seizures, convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose
* History of asthma, thyroidectomy, angioedema, severe liver, kidney, or cardiovascular disease, diabetes mellitus that can not be controlled by stable doses of insulin, or malignancy;
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy;
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* Acute diseases or acute stage of chronic diseases or use of antipyretic, analgesic drugs (eg: acetaminophen, ibuprofen, aspirin, etc.) and anti-allergic drugs (such as: loratadine, cetirizine, etc.) within 3 days preceding the vaccination;
* Untreated/uncontrolled hypertension before vaccination (16-17 years of age > 120 mmHg and / or diastolic blood pressure > 80 mmHg; 18-26 years of age with physical examination systolic blood pressure ≥140 mmHg and / or diastolic blood pressure ≥90 mmHg);
* Subjects who received whole blood, plasma, or immunoglobulin therapy within 3 months prior to vaccination;
* Received live attenuated vaccine within 28 days prior to vaccination;
* Received subunits or inactivated vaccines within 14 days prior to vaccination;
* Breastfeeding or pregnant, or within 6 weeks after the end of pregnancy;
* According to the judgment of the investigator, subjects who have any other factors that are not suitable for participating in this clinical trial.

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMT) of HPV neutralizing antibodies | 30 days postdose 3 (Month 7)
  HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 neutralizing antibodies GMT
Seroconversion Percentages to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 30 days postdose 3 (Month 7)
  Seroconversion is defined as a participant in PPS who was anti-HPV seronegative at Day 0 (before vaccination) and became seropositive 30days after the third dose (Month 7).

SECONDARY OUTCOMES:
Percentage of subjects reporting solicited local symptoms | 0-7 days after each dose
  Solicited local symptoms assessed including pain, redness, swelling, induration and pruritus.
Percentage of subjects reporting solicited general symptoms | 0-7 days after each dose
  Solicited general symptoms assessed including fever, headache, fatigue, nausea, diarrhea, vomiting, myalgia, allergic reaction
Percentage of subjects reporting unsolicited adverse events (AEs) | 0-30 days after each dose
  An unsolicited adverse event is defined as any adverse event (AE) reported in addition to those solicited during the clinical study.
Percentage of subjects reporting serious adverse events (SAEs) | Month 0 to Month 12
  Serious adverse events are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.

CONTACTS AND LOCATIONS:
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China